CLINICAL TRIAL: NCT06226558
Title: Prospective Observational Study of Asymptomatic cCMV Transmission to Infants for Virological Evaluation in New York State
Brief Title: Long-Term Outcomes of Children With Congenital CMV in New York State
Acronym: PROACTIVE NYS
Status: Recruiting | Type: Observational
Sponsor: Stony Brook University (Other)
Collaborators: Frontier Science & Technology Research Foundation, Inc. (Industry)
Responsible Party: Principal Investigator, Andrew S Handel, Physician, Stony Brook University
Other Study IDs: 75N94021D00018-75N94023F00001
Record Dates: First submitted 2023-12-19; First posted 2024-01-26 (Actual); Last update posted 2025-05-13 (Actual); Status verified 2025-05

CONDITIONS: Congenital CMV Infection; Sensorineural Hearing Loss
Keywords: Congenital CMV; cCMV; Congenital infection; Sensorineural hearing loss; SNHL
MeSH Terms: conditions — Cytomegalovirus Infections; Hearing Loss, Sensorineural

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 2 Years
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (4):
- Category 1: Confirmed cCMV infection identified by NYS newborn screen: Infants who have both a positive cCMV NYS newborn screen AND are positive for cCMV on confirmatory testing
- Category 2: Confirmed cCMV infection NOT identified by NYS newborn screen: Infants who have both a NEGATIVE cCMV NYS newborn screen AND are found to have cCMV on confirmatory testing
- Category 3: False-positive cCMV NYS newborn screen: Infants who have both a positive cCMV NYS newborn screen AND are NEGATIVE for cCMV on confirmatory testing
- Category 4: Premature infants with confirmed CMV infection on late positive NBS: Infants who are: (a) born prior to 37 weeks gestation AND (b) cCMV positive on any NYS newborn screen collected prior to 44 weeks gestational age AND (c) Have a positive cCMV confirmatory test obtained within 14 days of a positive NYS newborn screen

SUMMARY:
PROACTIVE NYS is a long-term follow-up study of all infants who test positive for congenital Cytomegalovirus infection (CMV) throughout New York State on the Newborn Screen. By following all infants who screen positive, we will learn important information about the range of symptoms caused by congenital CMV, from those babies with more severe findings to those with no symptoms.

In particular, our study will provide new information about many facets of congenital CMV, including:

* Developmental, hearing, neurologic, and vision outcomes
* The spectrum and timing of symptoms
* The impact congenital CMV has on the baby and its family
* How many babies are infected with congenital CMV in New York State How antiviral medications and other interventions impact outcomes of children with congenital CMV

Throughout the duration of the study, children will undergo routine developmental and hearing assessments, which will assist with early diagnosis of any infection complications.

Any child found to have a neurodevelopmental, hearing, or vision abnormality will be referred for appropriate evaluation and treatment.

Families will also be asked to complete periodic surveys about their experience with congenital CMV, both as a medical diagnosis and as it affects their day-to-day activities.

ELIGIBILITY:
Inclusion Criteria:

* Neonates born in New York State during cCMV NBS Pilot Program (September 27, 2023 - October 1, 2024)
* cCMV evaluation provided by a designated NYS cCMV clinical referral site
* Family willing and able to complete all study procedures
* Study participants meet criteria for one of the following four categories:
* 1. Category 1 (Confirmed cCMV identified by NBS Program): cCMV NYS newborn screen positive AND cCMV confirmatory test positive
* 2. Category 2 (Confirmed cCMV not identified by NBS Program): cCMV NYS newborn screen negative AND cCMV confirmatory test positive
* 3. Category 3 (False-positive cCMV screen): cCMV NYS newborn screen positive AND negative cCMV confirmatory test
* 4. Category 4 (Premature infants with confirmed CMV infection on late positive NBS): Infant born prior to 37 weeks gestation AND cCMV positive on any NYS newborn screen collected prior to 44 weeks gestational age AND Positive cCMV confirmatory test obtained within 14 days of a positive NBS

Exclusion Criteria:

* Neonate whose parents refuse participation in the long-term follow-up study

Ages: 0 Days to 1 Year | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: All infants referred by the New York State Newborn Screen Program to a clinical care referral site for a positive congenital CMV test will be approached for enrollment in PROACTIVE NYS. In addition, infants who are identified with cCMV as part of routine clinical care during the study period will be eligible to enroll in PROACTIVE NYS.
Sampling Method: Non-Probability Sample
Enrollment: 1000 (Estimated)
Dates: Start 2024-02-01 (Actual); Primary Completion 2025-10-01 (Estimated); Study Completion 2026-10-01 (Estimated)

PRIMARY OUTCOMES:
Congenital CMV infection rate | Study initiation to 1 year time point
  To determine the rate of confirmed congenital CMV in a statewide cohort

SECONDARY OUTCOMES:
cCMV neonatal sensorineural hearing loss | Through 4 weeks old
  Rate of neonatal sensorineural hearing decibel loss as determined by Auditory Brainstem Response testing
cCMV antiviral therapy utilization | 2 years
  Frequency of antiviral prescriptions
cCMV acquired sensorineural hearing loss | 2 years
  Rate of acquired sensorineural hearing decibel loss as determined by Auditory Brainstem Response testing
cCMV neurodevelopmental outcomes | 2 years
  Neurodevelopmental abnormalities as measured by Bayley Scales of Infant & Toddler Development-III.
  The Bayley-III includes Cognitive, Language, Motor, Social-Emotional, and Adaptive Behavior scales. Age-normalized scores are calculated for each domain, with a lower score indicating greater impairment.
cCMV-related quality of life | 2 years
  Quality of life score as determined by the Pediatric Quality of Life Inventory Infant Scales (PedsQL).
  The PedsQL Infant Scales consist of parent-reported psychosocial health symptoms. A higher score on the PedsQL indicates more severe psychosocial health symptoms.

CONTACTS AND LOCATIONS:
Locations (1):
- Stony Brook Children's Hospital, Stony Brook, New York, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Pesch MH, Saunders NA, Abdelnabi S. Cytomegalovirus Infection in Pregnancy: Prevention, Presentation, Management and Neonatal Outcomes. J Midwifery Womens Health. 2021 May;66(3):397-402. doi: 10.1111/jmwh.13228. Epub 2021 May 24. PMID 34031974
- [Background] Rawlinson WD, Boppana SB, Fowler KB, Kimberlin DW, Lazzarotto T, Alain S, Daly K, Doutre S, Gibson L, Giles ML, Greenlee J, Hamilton ST, Harrison GJ, Hui L, Jones CA, Palasanthiran P, Schleiss MR, Shand AW, van Zuylen WJ. Congenital cytomegalovirus infection in pregnancy and the neonate: consensus recommendations for prevention, diagnosis, and therapy. Lancet Infect Dis. 2017 Jun;17(6):e177-e188. doi: 10.1016/S1473-3099(17)30143-3. Epub 2017 Mar 11. PMID 28291720
- [Background] Fowler KB, Boppana SB. Congenital cytomegalovirus infection. Semin Perinatol. 2018 Apr;42(3):149-154. doi: 10.1053/j.semperi.2018.02.002. Epub 2018 Mar 2. PMID 29503048
- See also: PROACTIVE NYS Website — https://www.proactivenys.org/

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2023-10-25): https://cdn.clinicaltrials.gov/large-docs/58/NCT06226558/Prot_SAP_000.pdf
  • Informed Consent Form (2023-11-16): https://cdn.clinicaltrials.gov/large-docs/58/NCT06226558/ICF_001.pdf